CLINICAL TRIAL: NCT04062149
Title: Does Working on Single Leg Stance (SLS) Alongside Usual Physiotherapy Treatment Lead to a More Efficient Gait Pattern as Measured by the 10m Walk Test (10MWT) Compared to Those Receiving Usual Physiotherapy Only in Adults With Acquired Brain Injury? An Exploratory Study.
Brief Title: Does Improved Ability to Achieve Single Leg Stance Lead to a More Efficient Gait Pattern in Adults With Acquired Brain Injury?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Salford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B00678
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Acquired Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Exploratory pre-test - post-test experimental design
Who Masked: Participant
Masking Description: Participants will not know if thy have been allocated to the control or experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will be the group where the participants receive only their normal physiotherapy treatment.
  Interventions: Other: Usual physiotherapy
- Experimental Group (Experimental): The experimental group will be the group where participants receive physiotherapy aimed at improving their ability to stand on their weaker leg alongside their normal physiotherapy treatment.
  Interventions: Other: single leg stance treatment

INTERVENTIONS:
Other: single leg stance treatment — SLS treatment following the neurodevelopmental treatment (NDT). SLS is the ability of one limb to support the body's weight in a standing position. In gait it is the foot being in contact with the ground whilst the body passes over it and this stance phase of gait accounts for 60% of the gait cycle. The treatment approach of NDT has been chosen as this is the most common physiotherapy treatment option in the UK and is the most common option in the studies above. NDT is a problem-solving approach to the assessment and treatment of individuals with disturbances of function, movement and postural control due to a lesion of the central nervous system and provides an outline of the treatment required to achieve SLS which will form the basis of the intervention of this study.
  Arms: Experimental Group
Other: Usual physiotherapy — Individualised physiotherapy treatment approach, as per standard protocol, but it will not work specifically on SLS. Will be based on the neuro-developmental technique.
  Arms: Control Group

SUMMARY:
The purpose of the study is to see if a person can stand better on their weaker leg does this improve their walking ability following treatment specifically aimed at standing on leg. This will be compared to people who receive normal physiotherapy treatment not treatment specifically focusing on their ability to stand on their weaker leg. The study is being carried out as part of the researcher's Masters Degree. Participants will be allocated to either the control group (normal physiotherapy treatment) or the experimental group (normal physiotherapy plus physiotherapy working specifically on standing on the weaker leg). There is currently some evidence to show that working specifically on standing on one leg can improve a person's walking but this evidence is limited. Consequently, further research is warranted to identify any links between this treatment approach and walking ability.

DETAILED DESCRIPTION:
Acquired brain injury (ABI) incidence is 369 per 100,000 people internationally and 260 per 100,000 in the UK resulting in more than 900,000 people living with the long term effects of a cerebrovascular accident (CVA) and over 380,000 with impairments following traumatic brain injury. The ABI population often experience long term health problems affecting physical functioning, cognition, communication, emotion and behaviour with a loss of physical functioning and an inability to walk highlighted as the most negative aspect by patients. Several studies have identified people with neurological impairment who regain walking often mobilise at slower speeds with a mean gait velocity of 73.07cm/s for CVA survivors (60cm/s slower than healthy adults).

The gait cycle is described as having two major components, stance and swing phase. Stance has been determined as a pre-requisite for gait and a literature review found reduced stance ability correlates with gait abnormalities in CVA survivors. Consequently, given that a stronger and longer stance phase leads to a better swing phase and stance accounts for 60% of the gait cycle, stance can be considered the most important part of the gait cycle.

A person's ability to achieve SLS can be measured using the SLS test which assesses the time a person can stand on one leg. SLS test has excellent intra-rater reliability with an intraclass correlation coefficient (ICC) of 0.83 and excellent validity with a correlation of <10 seconds being a high predictor of mobility impairments for people with ABI. There is currently no definitive minimal clinical important difference (MCID) for the SLS test - current literature varies from 5.5 - 16.0 seconds - but as this study will assess the quality of each person's SLS test as opposed to the time the results will still be clinically relevant.

Goal Attainment Scale (GAS) based on the single leg stance (SLS) test will be used to assess quality as it is responsive to change, person-specific and quantitative, able to assess treatment interventions at the impairment and functional level, and is suitable for assessing and evaluating patient outcomes in the ABI population and is frequently used within neuro-rehabilitation. GAS has excellent intra-rater reliability (ICC 0.88-0.93) and inter-rater reliability (ICC 0.95) with good concurrent and predictive and moderate to good content and construct validity (r=0.28-0.63) across the ABI population.

The ten metre walk test (10MWT) will be used to assess gait efficiency. The 10MWT requires a patient to walk ten metres at a comfortable speed and the time taken to cover that distance is measured. Studies have found a relationship between reduced SLS and reduced speed in the 10MWT with improvements in gait speed demonstrated following intervention based on SLS. It is also hypothesised that increased gait speed results in a more efficient and fluent gait pattern. Consequently, 10MWT will be used in this study to demonstrate gait velocity and efficiency improvements. 10MWT is also one of the most common, reliable, efficient and robust outcomes measures within neuro-rehabilitation. 10MWT demonstrates excellent test-retest reliability (ICC 0.95-0.99) and excellent intra-rater (ICC 0.87-0.98) and inter-rater reliability (ICC 0.99). 10MWT also has excellent criterion validity of r=0.76-0.78 and excellent construct validity (r=0.62-0.92) for various outcome measures within the ABI population with an MCID of 0.14-0.16m/s.

Consequently, ABI results in a reduced ability to achieve SLS which has a negative influence on gait speed and efficiency. Studies of predominantly small samples have demonstrated working on SLS can improve gait speed and efficiency in CVA survivors and to a lesser extent the traumatic brain injury (TBI) population meaning there is a gap in the research surrounding the ABI population as a whole including TBI. Therefore, this study will aim to answer the question 'does improved ability to achieve SLS lead to a more efficient gait pattern in adults with acquired brain injury?' The null hypothesis is 'improved ability to achieve SLS does not lead to a more efficient gait pattern in patients with ABI'. The experimental hypothesis is 'improved ability to achieve SLS does lead to a more efficient gait pattern in patients with ABI'. This is a two-tailed hypothesis due to limited evidence regarding the testing direction.

This will be an exploratory pre-test - post-test experimental design as it allows testing of two variables (dependent and independent) to identify the cause and effect of specific events. This research design also helps determine if the subjects' performance is better, worse or unchanged and the inclusion of a control group will provide more convincing evidence of success or failure of treatment. The control group will receive an individualised physiotherapy treatment approach, but it will not work specifically on SLS i.e. they will receive their normal physiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ABI as diagnosed by a doctor following a brain scan
* Adults aged eighteen years or over
* Patients can be male or female
* Mobile >10m with or without assistance/walking aid
* Willing and able to provide written informed consent and scores >5 on orientation on FIM+FAM (FIM+FAM is an outcome measure used in all neuro-rehabilitation units in England, consequently, these data are already captured by the unit)
* Medically stable - able to fully take part in regular therapy - as determined by the unit's medical team

Exclusion Criteria:

* Diagnosed with a progressive neurological condition by a doctor
* Below eighteen years of age
* Mobile <10m or not mobile
* Unable or unwilling to give informed consent or scores <5 on orientation on FIM+FAM Medically unwell

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved gait speed as measured by an increase in metres per second in the 10m walk test (10MWT) | 6 weeks
  The 10m walk test (10MWT) is a measure of gait speed. Time to walk 10m is converted to metres/second. This will be completed pre and post intervention and the difference compared. An increase in speed (metres per second) demonstrates a positive outcome. A change of greater than 0.14m/s indicates a clinical important difference.

SECONDARY OUTCOMES:
Number of participants who improve their ability to achieve single leg stance (SLS) with a change in Goal Attainment Scale (GAS) T-score of greater than 10 | 6 weeks
  Goal Attainment Scale (GAS) enables patient outcomes to be documented on a scale of -2 to +2 with -1 accepted as the baseline and 0 as the anticipated outcome. This is completed pre and post intervention and converted to a T-score with a mean of 50. An increase in the T-score indicates a positive outcome. A difference of 10 is seen as a clinically important difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Trafford General Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen JL, Kautz SA, Neptune RR. Step length asymmetry is representative of compensatory mechanisms used in post-stroke hemiparetic walking. Gait Posture. 2011 Apr;33(4):538-43. doi: 10.1016/j.gaitpost.2011.01.004. Epub 2011 Feb 11. PMID 21316240
- [Background] Baker JM. Gait Disorders. Am J Med. 2018 Jun;131(6):602-607. doi: 10.1016/j.amjmed.2017.11.051. Epub 2017 Dec 27. PMID 29288631
- [Background] Brandstater ME, de Bruin H, Gowland C, Clark BM. Hemiplegic gait: analysis of temporal variables. Arch Phys Med Rehabil. 1983 Dec;64(12):583-7. PMID 6661021
- [Background] Bonora G, Mancini M, Carpinella I, Chiari L, Ferrarin M, Nutt JG, Horak FB. Investigation of Anticipatory Postural Adjustments during One-Leg Stance Using Inertial Sensors: Evidence from Subjects with Parkinsonism. Front Neurol. 2017 Jul 25;8:361. doi: 10.3389/fneur.2017.00361. eCollection 2017. PMID 28790972
- [Background] Bovend'Eerdt TJ, Dawes H, Izadi H, Wade DT. Agreement between two different scoring procedures for goal attainment scaling is low. J Rehabil Med. 2011 Jan;43(1):46-9. doi: 10.2340/16501977-0624. PMID 21042701
- [Background] Brock K, Haase G, Rothacher G, Cotton S. Does physiotherapy based on the Bobath concept, in conjunction with a task practice, achieve greater improvement in walking ability in people with stroke compared to physiotherapy focused on structured task practice alone?: a pilot randomized controlled trial. Clin Rehabil. 2011 Oct;25(10):903-12. doi: 10.1177/0269215511406557. Epub 2011 Jul 25. PMID 21788266
- [Background] Burnfield JM, Buster TW, Goldman AJ, Corbridge LM, Harper-Hanigan K. Partial body weight support treadmill training speed influences paretic and non-paretic leg muscle activation, stride characteristics, and ratings of perceived exertion during acute stroke rehabilitation. Hum Mov Sci. 2016 Jun;47:16-28. doi: 10.1016/j.humov.2016.01.012. Epub 2016 Feb 1. PMID 26845732
- [Background] Carvalho C, Sunnerhagen KS, Willen C. Walking performance and muscle strength in the later stage poststroke: a nonlinear relationship. Arch Phys Med Rehabil. 2013 May;94(5):845-50. doi: 10.1016/j.apmr.2012.11.034. Epub 2012 Dec 3. PMID 23219614
- [Background] Chomiak T, Pereira FV, Hu B. The single-leg-stance test in Parkinson's disease. J Clin Med Res. 2015 Mar;7(3):182-5. doi: 10.14740/jocmr1878w. Epub 2014 Dec 29. PMID 25584104
- [Background] Dorsch S, Ada L, Canning CG, Al-Zharani M, Dean C. The strength of the ankle dorsiflexors has a significant contribution to walking speed in people who can walk independently after stroke: an observational study. Arch Phys Med Rehabil. 2012 Jun;93(6):1072-6. doi: 10.1016/j.apmr.2012.01.005. Epub 2012 Mar 29. PMID 22464738
- [Background] Drummond, A. (1998). Research methods for therapists. Cheltenham: Cheltenham : Stanley Thornes.
- [Background] Evans JJ. Goal setting during rehabilitation early and late after acquired brain injury. Curr Opin Neurol. 2012 Dec;25(6):651-5. doi: 10.1097/WCO.0b013e3283598f75. PMID 23007008
- [Background] Gatrell, S. (2006). The use of the Bobath Concept to facilitate single leg stance and the influence of this on gait in patients following stroke. Synapse, Spring, 11-15.
- [Background] Graham JE, Ostir GV, Kuo YF, Fisher SR, Ottenbacher KJ. Relationship between test methodology and mean velocity in timed walk tests: a review. Arch Phys Med Rehabil. 2008 May;89(5):865-72. doi: 10.1016/j.apmr.2007.11.029. PMID 18452733
- [Background] Hurn J, Kneebone I, Cropley M. Goal setting as an outcome measure: A systematic review. Clin Rehabil. 2006 Sep;20(9):756-72. doi: 10.1177/0269215506070793. PMID 17005500
- [Background] Jacobs JV, Horak FB, Tran VK, Nutt JG. Multiple balance tests improve the assessment of postural stability in subjects with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2006 Mar;77(3):322-6. doi: 10.1136/jnnp.2005.068742. PMID 16484639
- [Background] Jarnlo, G. & Nordell, E. (2003). Reliability of the modified figure of eight - a balance performance test for elderly women. Physiotherapy Theory and Practice, 19(1), 35-43
- [Background] Jonsdottir J, Cattaneo D. Reliability and validity of the dynamic gait index in persons with chronic stroke. Arch Phys Med Rehabil. 2007 Nov;88(11):1410-5. doi: 10.1016/j.apmr.2007.08.109. PMID 17964880
- [Background] Kamphuis JF, de Kam D, Geurts AC, Weerdesteyn V. Is weight-bearing asymmetry associated with postural instability after stroke? A systematic review. Stroke Res Treat. 2013;2013:692137. doi: 10.1155/2013/692137. Epub 2013 Apr 28. PMID 23738232
- [Background] Khan F, Pallant JF, Turner-Stokes L. Use of goal attainment scaling in inpatient rehabilitation for persons with multiple sclerosis. Arch Phys Med Rehabil. 2008 Apr;89(4):652-9. doi: 10.1016/j.apmr.2007.09.049. PMID 18373995
- [Background] King IM. King's theory of goal attainment in practice. Nurs Sci Q. 1997 Winter;10(4):180-5. doi: 10.1177/089431849701000411. PMID 9416120
- [Background] Krasny-Pacini A, Hiebel J, Pauly F, Godon S, Chevignard M. Goal attainment scaling in rehabilitation: a literature-based update. Ann Phys Rehabil Med. 2013 Apr;56(3):212-30. doi: 10.1016/j.rehab.2013.02.002. Epub 2013 Feb 28. PMID 23562111
- [Background] Korley FK, Diaz-Arrastia R, Falk HJ, Peters ME, Leoutsakos JS, Roy D, Rao V, Sair HI, Ofoche U, Hall AJ, Akbari F, Van Meter TE, Everett AD, Van Eyk JE, Bechtold KT. Prevalence of Incomplete Functional and Symptomatic Recovery among Patients with Head Injury but Brain Injury Debatable. J Neurotrauma. 2017 Apr 15;34(8):1531-1538. doi: 10.1089/neu.2016.4723. Epub 2016 Dec 20. PMID 27784200
- [Background] Lennon S. Physiotherapy practice in stroke rehabilitation: a survey. Disabil Rehabil. 2003 May 6;25(9):455-61. doi: 10.1080/0963828031000069744. PMID 12745940
- [Background] Lennon S, Ashburn A, Baxter D. Gait outcome following outpatient physiotherapy based on the Bobath concept in people post stroke. Disabil Rehabil. 2006 Jul 15-30;28(13-14):873-81. doi: 10.1080/09638280500535132. PMID 16777775
- [Background] Mar J, Arrospide A, Begiristain JM, Larranaga I, Elosegui E, Oliva-Moreno J. The impact of acquired brain damage in terms of epidemiology, economics and loss in quality of life. BMC Neurol. 2011 Apr 18;11:46. doi: 10.1186/1471-2377-11-46. PMID 21496356
- [Background] Morris M, Iansek R, Smithson F, Huxham F. Postural instability in Parkinson's disease: a comparison with and without a concurrent task. Gait Posture. 2000 Dec;12(3):205-16. doi: 10.1016/s0966-6362(00)00076-x. PMID 11154931
- [Background] Michielsen M, Vaughan-Graham J, Holland A, Magri A, Suzuki M. The Bobath concept - a model to illustrate clinical practice. Disabil Rehabil. 2019 Aug;41(17):2080-2092. doi: 10.1080/09638288.2017.1417496. Epub 2017 Dec 17. PMID 29250987
- [Background] Park YH, Kim YM, Lee BH. An ankle proprioceptive control program improves balance, gait ability of chronic stroke patients. J Phys Ther Sci. 2013 Oct;25(10):1321-4. doi: 10.1589/jpts.25.1321. Epub 2013 Nov 20. PMID 24259785
- [Background] Patterson KK, Gage WH, Brooks D, Black SE, McIlroy WE. Changes in gait symmetry and velocity after stroke: a cross-sectional study from weeks to years after stroke. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):783-90. doi: 10.1177/1545968310372091. Epub 2010 Sep 14. PMID 20841442
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Peters DM, Jain S, Liuzzo DM, Middleton A, Greene J, Blanck E, Sun S, Raman R, Fritz SL. Individuals with chronic traumatic brain injury improve walking speed and mobility with intensive mobility training. Arch Phys Med Rehabil. 2014 Aug;95(8):1454-60. doi: 10.1016/j.apmr.2014.04.006. Epub 2014 Apr 24. PMID 24769069
- [Background] Research methods for clinical therapists: applied project design and analysis Carolyn M Hicks Research methods for clinical therapists: applied project design and analysis Churchill LIvingstone 352 Fifth edition pound22.99 9780043074301 [Formula: see text]. Nurse Res. 2010 Oct 22;18(1):89. doi: 10.7748/nr.18.1.89.s3. PMID 27707351
- [Background] Raine, S., Meadows, L., & Lynch-Ellerington, M. (2009). The Bobath concept : theory and clinical practice in neurological rehabilitation. Chichester: Chichester : Wiley-Blackwell
- [Background] Ryan, S. (2014) Goal Attainment Scale. Retrieved from: https://www.sralab.org/rehabilitation-measures/goal-attainment-scale
- [Background] Ryan, S. (2014). 10m walk test. Retrieved from: https://www.sralab.org/rehabilitation-measures/10-meter-walk-test
- [Background] Ryan, S. (2013). Single leg stance or one-legged stance test. Retrieved from: https://www.sralab.org/rehabilitation-measures/single-leg-stance-or-one-legged-stance-test
- [Background] Schmid A, Duncan PW, Studenski S, Lai SM, Richards L, Perera S, Wu SS. Improvements in speed-based gait classifications are meaningful. Stroke. 2007 Jul;38(7):2096-100. doi: 10.1161/STROKEAHA.106.475921. Epub 2007 May 17. PMID 17510461
- [Background] Shankar, S., Marshall, S. & Zumbo, B. (2019). A systematic review of validation practices for the Goal Attainment Scaling Measure. Journal of Psychoeducational Assessment, 3(1), 1-20
- [Background] Sherrington C, Lord SR. Reliability of simple portable tests of physical performance in older people after hip fracture. Clin Rehabil. 2005 Aug;19(5):496-504. doi: 10.1191/0269215505cr833oa. PMID 16119405
- [Background] Shumway-Cook, A. (2007). Motor control : translating research into clinical practice (3rd ed. ed.). Philadelphia, PA ; London: Philadelphia, PA ; London : Lippincott Williams & Wilkins
- [Background] Skinner A, Turner-Stokes L. The use of standardized outcome measures in rehabilitation centres in the UK. Clin Rehabil. 2006 Jul;20(7):609-15. doi: 10.1191/0269215506cr981oa. PMID 16894804
- [Background] Smithson F, Morris ME, Iansek R. Performance on clinical tests of balance in Parkinson's disease. Phys Ther. 1998 Jun;78(6):577-92. doi: 10.1093/ptj/78.6.577. PMID 9626270
- [Background] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Background] Tyson S, Connell L. The psychometric properties and clinical utility of measures of walking and mobility in neurological conditions: a systematic review. Clin Rehabil. 2009 Nov;23(11):1018-33. doi: 10.1177/0269215509339004. Epub 2009 Sep 28. PMID 19786420
- [Background] Tilson JK, Sullivan KJ, Cen SY, Rose DK, Koradia CH, Azen SP, Duncan PW; Locomotor Experience Applied Post Stroke (LEAPS) Investigative Team. Meaningful gait speed improvement during the first 60 days poststroke: minimal clinically important difference. Phys Ther. 2010 Feb;90(2):196-208. doi: 10.2522/ptj.20090079. Epub 2009 Dec 18. PMID 20022995
- [Background] van Loo MA, Moseley AM, Bosman JM, de Bie RA, Hassett L. Test-re-test reliability of walking speed, step length and step width measurement after traumatic brain injury: a pilot study. Brain Inj. 2004 Oct;18(10):1041-8. doi: 10.1080/02699050410001672314. PMID 15370902
- [Background] Wade, D. T. (1992). Measurement in neurological rehabilitation. Oxford ; New York: Oxford ; New York : Oxford University Press.
- [Background] Wang P, Low KH, McGregor AH, Tow A. Detection of abnormal muscle activations during walking following spinal cord injury (SCI). Res Dev Disabil. 2013 Apr;34(4):1226-35. doi: 10.1016/j.ridd.2012.12.013. Epub 2013 Feb 6. PMID 23396198
- [Background] Watson, M. (2002). Refining the ten-metre walk test for use with neurologically impaired people. Physiotherapy, 88(7), 386-397
- [Background] Whittle, M. (2007). Gait analysis : an introduction (4th ed. ed.). Edinburgh: Edinburgh : Butterworth-Heinemann.
- [Background] Wolf SL, Catlin PA, Gage K, Gurucharri K, Robertson R, Stephen K. Establishing the reliability and validity of measurements of walking time using the Emory Functional Ambulation Profile. Phys Ther. 1999 Dec;79(12):1122-33. PMID 10630281